CLINICAL TRIAL: NCT05854264
Title: Lung Microbiota in Traumatic Brain Injury
Brief Title: Influence of Nutrition on Lung Microbiota in Traumatic Brain Injury
Acronym: Microbiota
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, Principal Investigator, University of Foggia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 46/CE/2022
Record Dates: First submitted 2023-04-22; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: specialized nutrition group
Who Masked: Participant
Masking Description: specialized nutrition and microbiota analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- microbiota and specialized nutrition (Active Comparator): microbiota analysis in lower lavage (Bronco Alveolar Lavage: BAL) samples in patietns treated with specialized nutrition
  Interventions: Dietary Supplement: specialized nutrition
- microbiota and standard nutrition (Sham Comparator): microbiota analysis in lower lavage (Bronco Alveolar Lavage: BAL) samples in patients treated with standard nutrition
  Interventions: Dietary Supplement: standard enteral nutrition

INTERVENTIONS:
Dietary Supplement: standard enteral nutrition — standard enteral nutrition. The calories (25 kcal/kg/die) and protein (1.2 g/kg/die) target will be progressively reached in the first week of ICU stay.
  Arms: microbiota and standard nutrition
Dietary Supplement: specialized nutrition — specialized enteral nutrition. The calories (25 kcal/kg/die) and protein (1.2 g/kg/die) target will be progressively reached in the first week of ICU stay.
  Arms: microbiota and specialized nutrition

SUMMARY:
Role of immunonutrition in modulating the lung microbiota of intubated TBJ patients and how this interaction may affect the infections and outcomes.

For these reasons, the aims of our study are the evaluation of the impact of immunonutrition on the lung microbiota and the relationship between lung microbiota and infection in TBJ patients in ICU.

DETAILED DESCRIPTION:
Traumatic brain injury patients, requiring mechanical ventilation admitted to ICU will be randomly divide in two groups receiving standard nutrition or specialized formula.

Lower lavage (Bronco Alveolar Lavage: BAL) samples will be collected at admission in ICU and at day 7 for the microbiota analysis. Clinical follow-up at day 28 will be obtained

ELIGIBILITY:
Inclusion Criteria:

* adults (age > 18 years),
* paziente with traumatic brain injury

Exclusion Criteria:

* pregnant women,
* patients with gastric content inhalation
* patients with chronic inflammatory bowel diseases
* patients underwent major abdominal surgery and/or organs/tissues transplant
* patients on corticosteroid and/or immunosuppressive therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
infection | pulmonary infection within 28 days
  pulmonary infection in mechanically ventilated patients

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedali Riuniti, Foggia, Apulia, Italy